CLINICAL TRIAL: NCT02722434
Title: MC15C1 Randomized Scrambler Therapy vs TENS for the Treatment of Chemotherapy-Induced Peripheral Neuropathy
Brief Title: MC5-A Scrambler Therapy or TENS Therapy in Treating Patients With Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC15C1; NCI-2016-00368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC15C1 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-06

CONDITIONS: Pain; Peripheral Neuropathy; Tingling
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases; Paresthesia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (MC5-A scrambler therapy) (Experimental): Patients undergo MC5-A scrambler therapy over 30 minutes for 10 consecutive weekdays.
  Interventions: Other: Laboratory Biomarker Analysis; Other: MC5-A Scrambler Therapy; Other: Questionnaire Administration
- Arm II (TENS therapy) (Active Comparator): Patients undergo TENS therapy over 30 minutes daily for 14 days.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: MC5-A Scrambler Therapy — Undergo Scrambler therapy
  Other Names: Scrambler Therapy
  Arms: Arm I (MC5-A scrambler therapy)
Other: Questionnaire Administration — Ancillary studies
Other: Transcutaneous Electrical Nerve Stimulation — Undergo TENS
  Other Names: TENS; transcutaneous electric nerve stimulation
  Arms: Arm II (TENS therapy)

SUMMARY:
This randomized clinical trial studies how well MC5-A scrambler therapy or transcutaneous electrical nerve stimulation (TENS) therapy work in treating patients with chemotherapy-induced peripheral neuropathy (a nerve problem that causes pain, numbness, tingling, swelling, or muscle weakness in different parts of the body). MC5-A scrambler therapy is a type of treatment for nerve pain that uses electrodes placed on the skin, where electricity is carried from the electrodes through the skin and blocks the pain. TENS is a procedure in which mild electric currents are applied to some areas of the skin. It is not yet known whether TENS therapy is more effective than MC5-A scrambler therapy in treating chemotherapy-induced peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the efficacy of scrambler therapy (MC5-A scrambler therapy) compared to TENS therapy for pain and/or tingling related to chemotherapy-induced peripheral neuropathy (CIPN).

II. Evaluate the tolerability of scrambler therapy and compare it to TENS therapy, in this population.

III. Evaluate whether scrambler therapy, compared to TENS therapy, can decrease the use of pain medication for CIPN.

IV. Explore whether messenger ribonucleic acid (mRNA) gene expression before and after scrambler therapy shows similar findings to what Starkweather et al observed.

V. Utilizing high-field magnetic resonance imaging (MRI), to define alterations in functional differences (using resting state blood-oxygen-level dependent [BOLD] measures to measure differences in functional connectivity) in treated with the scrambler device in the setting of chemotherapy induced peripheral neuropathy pain.

VI. Explore whether scrambler therapy will alter sensation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo MC5-A scrambler therapy over 30 minutes for 10 consecutive weekdays.

ARM II: Patients undergo TENS therapy over 30 minutes daily for 14 days.

Patients in both Arms, may crossover to the opposite Arm for an additional 2 weeks of treatment if they elect.

After completion of study treatment, patients are followed up weekly for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pain or symptoms of CIPN of >= 3 months duration, for which the patient wants intervention

  * Note: neurotoxic chemotherapy must have been completed >= 3 months prior to registration and there must be no further planned neurotoxic chemotherapy for > 5 months after registration
* Patients have to relate that tingling or pain was at least a four out of ten problem =< 7 days prior to registration, on a 0-10 scale where zero was no problem and ten was the worst possible problem

  * Note: the patient is expected to have tingling or pain of at least 4/10 at the time of the first treatment
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 0, 1, or 2
* Life expectancy >= 6 months
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to provide informed written consent
* Case review by the study chair, or designate, as a case where treatment should be tried

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Existing operational implantable drug delivery systems, e.g. Medtronic Synchromed
* Existing implantable medical electronic devices, life-supporting medical devices, and medical monitoring devices

  * Note: metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed as are central venous access devices
* History of myocardial infarction or ischemic heart disease within the past six months
* History of epilepsy, brain damage, use of anticonvulsants for seizure prevention, concurrently using ketamine, symptomatic brain metastases
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study
* Currently receiving gabapentin or pregabalin and not willing to be weaned off of these medications prior to Scrambler therapy initiation

  * Note: it is OK to continue these medications in patients who are receiving TENS
* History of peripheral neuropathy prior to receiving neurotoxic chemotherapy
* Prior treatment with Scrambler therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Childs DS, Le-Rademacher JG, McMurray R, Bendel M, O'Neill C, Smith TJ, Loprinzi CL. Randomized Trial of Scrambler Therapy for Chemotherapy-Induced Peripheral Neuropathy: Crossover Analysis. J Pain Symptom Manage. 2021 Jun;61(6):1247-1253. doi: 10.1016/j.jpainsymman.2020.11.025. Epub 2020 Nov 27. PMID 33249081
- [Derived] Cathcart-Rake EJ, Hilliker DR, Loprinzi CL. Chemotherapy-induced neuropathy: Central resolution of a peripherally perceived problem? Cancer. 2017 Jun 1;123(11):1898-1900. doi: 10.1002/cncr.30650. Epub 2017 Mar 3. No abstract available. PMID 28257145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
Started (Registered/Randomized) | 25 | 25
Started Treatment | 24 | 25
Completed (Completed Treatment) | 24 | 22
Not Completed | 1 | 3
Not completed — Withdrawal Prior to Beginning Treatment | 1 | 0
Not completed — Withdrawal After Beginning Treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: All Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 61.0 [30.0 to 82.0] | 61.0 [52.0 to 77.0] | 61.0 [30.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 21 | 24 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 15 | 14 | 29
    1 | 9 | 10 | 19
    2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve at Least a 50% Reduction in Their Primary Problematic Symptom (Either Pain or Tingling) From Baseline on Day 14
Description: The number of participants who achieve at least a 50% reduction in their primary problematic symptom (either pain or tingling) from baseline on Day 14. The participant specified their primary problematic symptom (either pain or tingling) and primary problematic area (either upper or lower extremity) at registration; the respective items used to measure each symptom are considered for this outcome measure. Pain and tingling are measured using either item #6 (How much tingling have you had in your [fingers or hands; toes or feet] on average over the past 24 hours?) or item #9 (How much pain have you had in your [fingers or hands; toes or feet] on average over the past 24 hours?). Both items use the same scale: 0=None, 10=As bad as can be, with higher scores indicating worse outcome on either the Patient Questionnaire: Before Each Treatment for Upper Extremity Neuropathy or Patient Questionnaire: Before Each Treatment for Lower Extremity Neuropathy at baseline and Day 14.
Time Frame: Baseline to Day 14
Population: All Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
Number analyzed (Participants) | 25 | 25
Participants | 10 | 5
Statistical Analysis 1: Comparison: Arm I (MC5-A Scrambler Therapy) vs Arm II (TENS Therapy); Test type: Superiority; p = 0.1228, Chi-squared

2. Secondary Outcome: Number of Participants Indicating Yes, No, or Unsure for Therapy Recommendation to Other Patients With Similar Problems on the Subjective Global Impression of Change Instrument
Description: The number of participants indicating 'Yes' for 'Therapy recommendation to other patients with similar problems' on the Subjective Global Impression of Change (SGIC) instrument. The SGIC questionnaire is used to assess the change in quality of life.
Time Frame: At 10 weeks
Population: Participants who completed the SGIC 'Therapy recommendation to other patients with similar problems' item at Week 10 are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
Number analyzed (Participants) | 21 | 17
Participants
  Yes | 16 | 7
  No | 0 | 7
  Unsure | 5 | 3
Statistical Analysis 1: Comparison: Arm I (MC5-A Scrambler Therapy) vs Arm II (TENS Therapy); Test type: Superiority; p = 0.004, Fisher Exact

3. Secondary Outcome: Change in Sensory, Motor, and Autonomic Neuropathy Subscale Scores From Baseline to Week 10
Description: The change in Sensory, Motor, and Autonomic Neuropathy Subscale Scores from Baseline to Week 10 will be derived by subtracting the baseline score from the scores at Week 10. The European Organisation for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ CIPN-20) Instrument contains 20 items assessing sensory (9 items), motor (8 items), and autonomic symptoms (3 items), using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"). The range of change in subscale scores is -3 to 3. With a total range for sensory being -27 to 27 and motor being -24 to 24 and autonomic being -9 to 9. With negatives meaning a decrease in neuropathy and positive being an increase.
Time Frame: Up to 10 weeks
Population: Participants who completed all subscale items from the EORTC QLQ CIPN-20 at baseline and Week 10 are included in this analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
Number analyzed (Participants) | 25 | 25
score on a scale
  Sensory Subscale: number analyzed (Participants) | 21 | 16
  Sensory Subscale | -0.4 [-2.4 to 0.1] | -0.6 [-1.4 to 0.3]
  Motor Subscale: number analyzed (Participants) | 22 | 17
  Motor Subscale | -0.1 [-1.5 to 0.5] | -0.3 [-1.7 to 0.3]
  Autonomic Subscale: number analyzed (Participants) | 22 | 17
  Autonomic Subscale | 0.0 [-1.0 to 0.3] | 0.0 [-1.0 to 0.5]
Statistical Analysis 1: Comparison: Arm I (MC5-A Scrambler Therapy) vs Arm II (TENS Therapy); Sensory Subscale; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (MC5-A Scrambler Therapy) vs Arm II (TENS Therapy); Motor Subscale; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm I (MC5-A Scrambler Therapy) vs Arm II (TENS Therapy); Autonomic Subscale; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants Using Acetaminophen as Pain Medication
Description: The number of participants using acetaminophen as pain medication is reported below.
Time Frame: Up to 10 weeks
Population: All Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
Number analyzed (Participants) | 25 | 25
Participants | 8 | 9

5. Other Pre Specified Outcome: Change in mRNA Gene Expression
Description: In a descriptive manner, the gene expression will be compared to what was previously reported by Starkweather et al.
Time Frame: Baseline to up to 10 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Functional MRI (fMRI)
Description: Changes in fMRI following Scrambler therapy will be described in the subset of patients selected for this component of the study.
Time Frame: Baseline to up to 10 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Sensation
Description: Descriptive statistics will be used for the data from Quantitative Sensory Testing.
Time Frame: Baseline to up to 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: Participants who completed the study and did not withdraw prior to starting treatment are evaluable for adverse events.
Arm/Group | Arm I (MC5-A Scrambler Therapy) | Arm II (TENS Therapy)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MC5-A Scrambler Therapy) (N=24) | Arm II (TENS Therapy) (N=25)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT02722434/Prot_SAP_000.pdf